CLINICAL TRIAL: NCT01642810
Title: Online Acceptance-Based Behavioural Treatment for Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Heather Simister, PhD Candidate, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2012:179
Record Dates: First submitted 2012-06-25; First posted 2012-07-17 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Fibromyalgia Syndrome
Keywords: Online treatment for Fibromyalgia Syndrome; Acceptance-based behavioural treatment
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment-as-usual (Active Comparator): Participants continue their pre-study treatment plan, based on their physician/other professional recommendations
  Interventions: Other: Will vary per participant
- Online ABBT treatment + TAU (Experimental): Participants to complete a 6-unit online Acceptance-based behavioural treatment including training in pacing, mindfulness, acceptance, cognitive defusion, willingness, and exercise while also maintaining their pre-study treatment.
  Interventions: Behavioral: Acceptance-based behavioural therapy; Other: Will vary per participant

INTERVENTIONS:
Behavioral: Acceptance-based behavioural therapy — Behavioral intervention focusing on acceptance, mindfulness and values-based living instead of focus on symptom control
  Arms: Online ABBT treatment + TAU
Other: Will vary per participant — Participants will continue pre-study treatment under their current licensed practitioners. Intervention may include drug treatment, physical therapy, or other

SUMMARY:
A recent study published by the Canadian Pain Society estimated the direct health care costs of chronic pain to be about 6 billion dollars. Over 1/3 of all Canadians reported that they either missed work or experienced reduced productivity due to chronic pain. Fibromyalgia Syndrome (FMS)is a condition that affects up to 10% of the Canadian population, many of whom are still in the prime of their lives. While pain and fatigue are prominent symptoms, FMS sufferers often experience sleep disturbance, gastrointestinal upset, chronic headache, memory and thinking problems, and depression. Standard treatments focus on medication and physical exercise but are not always successful. Acceptance-Based behavioural therapy (ABBT) is a relatively new approach that has been effective not only in treating mental health concerns such as anxiety and depression, but also other medical conditions such as diabetes and chronic pain. A novel ABBT for FMS was developed and pilot tested with a small group of participants. The results of this preliminary study were promising. Unfortunately, many people cannot adequately access available treatment due to long wait lists, prohibitive costs, or time/location constraints. Online treatments may offer improved access to care without reducing the effectiveness of treatment. Therefore, the ABBT for FMS used in the pilot study is being adapted to an online format and will be evaluated with a larger group of participants. A wait-list/control group will be employed to evaluate the effectiveness of the online treatment as compared with treatment-as-usual. If found effective, this treatment would offer patients easier access to care at a significantly reduced cost to the health care system.

DETAILED DESCRIPTION:
The current study extended a pilot study (Shay, Tkachuk, Simister, Bailly, & Skrabek, 2011), modifying the previous treatment to a 6 unit program that could be delivered online. Sixty-one participants completed the study, being randomly assigned to an online ABBT plus treatment-as-usual (online ABBT + TAU) group or a treatment-as-usual alone (TAU) group. All participants completed a series of self-report measures at baseline, at post-treatment, and at a 3-month follow-up. Linear mixed modelling supported significant differences between the groups in favour of the ABBT + TAU treatment group on the primary outcome measure (Fibromyalgia Impact Questionnaire-Revised (FIQ-R); F (2, 52.82) = 20.10, p < .0001) following treatment. The online ABBT + TAU group also had significantly greater improvements in depression, pain, acceptance, perceived helplessness, and kinesiophobia. Increased acceptance mediated the effects of treatment on improvements in FMS quality of life and FMS impact, while reduced helplessness mediated the effects of treatment on improvements in level of reported pain. Comments and subjective ratings of improvement were consistent with the quantitative results. Participants rated mindfulness (contact with present moment experience) as the most useful treatment unit.

ELIGIBILITY:
Inclusion Criteria:

* Participants of either sex aged 18 years and older with a formal diagnosis of FMS will be recruited.
* Individuals younger than 18 years of age will be excluded in order to ensure all participants have reached the age of majority and can provide consent.
* They will have a pain intensity rating of at least 4/10 based on self-report. Participants will also be screened using the Wolfe et al (2010) criteria during the in-person session to ensure they meet criteria for FMS.
* Must reside in and complete study from within Manitoba, Canada

Exclusion Criteria:

* People with co-morbidities such as rheumatologic conditions, other conditions affecting the immune system (e.g. chronic fatigue syndrome, multiple sclerosis, lupus), brain injury, cognitive impairment that would limit a participant's ability to complete informed consent, active psychosis, substance abuse, uncontrolled major depression or bipolar disorder, active suicidality, or those who have current active injury claims will be excluded.
* Given the use of a large amount of reading materials, participants will be asked if they have completed at least grade 9 in high school. Those who have only completed grade 8 or lower will be excluded.
* Further, participants will be asked to maintain their pre-study treatment regime and not making changes to their medications or beginning other treatments for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Fibromyalgia Impact Questionnaire-revised | baseline, 2 months, 5 months
  Assesses overall impact of Fibromyalgia symptoms on daily functioning

SECONDARY OUTCOMES:
Change from baseline in Center for Epidemiological Studies Depression Scale | Baseline, 2 months, 5 months
  Evaluation of depressive symptoms
Change from baseline in Chronic Pain Acceptance Questionnaire | Baseline, 2 months, 5 months
  Overall acceptance of chronic pain
Change from baseline in Cognitive Fusion Questionnaire | Baseline, 2 months, 5 months
  Evaluation of fusion with thoughts
Change from baseline in McGill Pain Questionnaire- short form | Baseline, 2 months, 5 months
  subjective measure of type and severity of pain
Change from baseline in Five Facet Mindfulness Questionnaire | Baseline, 2 months, 5 months
  Measure of mindfulness skills
Change from baseline in Pittsburgh Sleep Quality Index | Baseline, 2 months, 5 months
  Measure of sleep quality and quantity
Change from baseline in Tampa Scale of Kinesiophobia-11 | Baseline, 2 months, 5 months
  Measure of fear of movement
Change from baseline in Valued Living Questionnaire | Baseline, 2 months, 5 months
  Measure of values, and how consistently one lives those values
Global Assessment Scale | 2 months
  unpublished scale evaluating the impact of treatment on symptoms, and how useful participants found the treatment protocol

CONTACTS AND LOCATIONS:
Overall Officials: Heather Simister, MA, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada